CLINICAL TRIAL: NCT02398435
Title: Open-label, Multicenter, Dose-escalating Phase II Study to Investigate the Safety, Tolerability, and Early Signs of Efficacy of Subcutaneous Administrations of Tadekinig Alfa (IL-18BP) in Patients With Adult -Onset Still's Disease (AoSD) During 12 Weeks
Brief Title: Therapeutic Use of Tadekinig Alfa in Adult-onset Still's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AB2 Bio Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AOSD-2014-001
Record Dates: First submitted 2015-02-23; First posted 2015-03-25 (Estimated); Last update posted 2016-12-06 (Estimated); Status verified 2016-08

CONDITIONS: Still's Disease, Adult-Onset
Keywords: Auto-inflammatory disease; Still's disease; Arthritis Rheumatoid; IL-18; interleukin-18; IL-18 binding protein
MeSH Terms: conditions — Still's Disease, Adult-Onset; Arthritis, Juvenile; Arthritis, Rheumatoid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cohort 80 mg (Experimental): Cohort 1 included 10 patients. Patients received Tadekinig alfa s.c with a dosage of 80mg. Safety assessments were conducted by data safety monitoring board. Non-responder patients were upscaled to next dose (160mg) after 3 weeks of treatment.
  Interventions: Biological: Tadekinig alfa (recombinant human IL-18 binding protein)
- Cohort 160 mg (Experimental): Cohort 2 included 13 patients. all patients were treated with Tadekinig alfa s.c with a dosage of 160mg. Safety was evaluated by data safety monitoring board.
  Interventions: Biological: Tadekinig alfa (recombinant human IL-18 binding protein)

INTERVENTIONS:
Biological: Tadekinig alfa (recombinant human IL-18 binding protein) — Patients received the study treatment three times a week subcutaneously.

SUMMARY:
The objective of this study is to assess safety, tolerability and early signs of efficacy of the investigational drug Tadekinig alfa in Adult-onset Still's disease, a rare polygenic auto-inflammatory disorder for which treatment remains empirical.

This disease is characterized by a daily spiking fever, arthralgia / arthritis, and skin rashes with frequent components of sore throat, lymphadenopathies and neutrophilic leukocytosis. The etiology is unknown. In addition to the above-mentioned clinical features, the diagnosis includes some laboratory components that reflect the systemic inflammation: high erythro-sedimentation rate, C-reactive protein, high serum ferritin and high levels of interleukin 18 (IL-18).

Tadekinig alfa is the drug name for recombinant human interleukin-18 binding protein (IL-18BP). This investigational drug was tested in healthy volunteers, psoriasis and rheumatoid arthritis patients in phase I studies. It demonstrated good safety and tolerability profile with only mild adverse events in the injection site.

DETAILED DESCRIPTION:
The hypothesis of this study considers high levels of IL-18 during active Adult-onset still's disease as the therapeutic target. Treatment with IL-18BP will permit to inhibit the pro-inflammatory cascade triggered by IL-18 and may help to manage the different components of the disease.

This study is an open label, dose-finding study involving multiple centers in Europe. Two dose cohorts (80mg and 160mg) were treated during twelve weeks and followed-up for four more weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years and older, diagnosed as AoSD based on the presence of the Yamaguchi criteria with active disease (see appendix 2), irrespective of the continuation of the permitted treatment mentioned below
* Patients with active disease will be considered if they exhibit at least two of the Yamaguchi's major criteria (see appendix 2) at the screening visit plus at least either fever or elevation of markers of inflammation (CRP ≥ 10 mg/L).
* Patients that have been exposed to NSAIDS, Prednisone (at least 5mg/day for ≥1 month) and/or synthetic sDMARDs (methotrexate at a dose of at least 10mg/day for ≥ 3 months) without response to treatment or with incomplete response to treatment
* Women of childbearing potential with negative pregnancy test at screening, V3, V4, V5 and V6 and that agree to follow highly effective birth control recommendations during the study and until 1 month after the end of the treatment. Birth control methods that are considered as highly effective are either: combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation, progestogen-only hormonal contraception associated with inhibition of ovulation, intrauterine device (IUD), intrauterine hormone-releasing system (IUS), bilateral tubal occlusion, vasectomized partner or sexual abstinence.

In each case of delayed menstrual period (over one month between menstruations, confirmation of absence of pregnancy is strongly recommended. This recommendation also applies to women of child bearing potential with infrequent or irregular menstrual cycles.

As regards the duration of contraception after the study, taking into account the median half-life of Tadekinig alfa of almost 40h, 5 half-lives represent duration of 200 hours. In order to be on the safe side, a post-study contraception duration of - Patients can maintain treatment with stable doses of Non-Steroidal anti-inflammatory Drugs (NSAIDs), Prednisone (stable dose of Prednisone of at least 5mg/day), and sDMARDs during Tadekinig alfa treatment (methotrexate at a dose of at least 10mg/week). Specifically baseline levels of prednisone treatment can be maintained or tapered (due to patient improvement), any requirement for prednisone increase during treatment will be considered a treatment failure.

* Ability to understand and willingness to sign a written informed consent
* Previous treatments with biologicals are allowed if the following wash-out periods are respected: one week for anakinra, two weeks for etanercept, and 6 weeks for, adalimumab, certolizumab, golimumab, tocilizumab, abatacept and 8 weeks for infliximab. Previous rituximab administration will require 6 months of washout and normal B-cell counts and previous treatment with canakinumab will require 6 months of washout.

Exclusion Criteria:

* Patients with a first episode of AoSD with less than one month of therapy with Prednisone or sDMARDs
* Patients with active or chronic infections (i.e. Tuberculosis (TB), HIV, HBV & HCV)
* Patients suffering from inherited immunodefinciency diseases
* Patients suffering from immune-mediated inflammatory diseases, including RA, SLE, etc. or spondylarthropathies, or inflammatory bowel disease.
* Patients with white blood cell counts below 2'500 cells/mm3
* Concomitantly treated with biologicals
* Women of childbearing potential who are unwilling to use highly effective birth control methods (see definition in Inclusion criteria above) up to 1 month after the end of her participation in the study.
* Inability to understand and unwilling to sign a written informed consent
* Any acute or chronic life-threatening disease: Such as cancer, and irreversible organ failures of heart, liver, lung and kidney (creatinine not higher than 1.5 X upper limit of normal).
* Patients having received adalimumab, certolizumab, golimumab, tocilizumab, abatacept within 6 weeks, infliximab within 8 weeks, canakinumab within 6 months, etanercept within 2 weeks, or anakinra 1 week prior to the start of Tadekinig alfa will not be enrolled into the study. Patients that have received rituximab within 6 months and/or have persistent low B-cell counts will not be eligible for enrolment.
* Subject who cannot be expected to comply with the study procedures
* Currently participating or having participated in another clinical trial during the last 4 weeks prior to the beginning of this study.
* Patients with no social security coverage
* Patients with a history of severe hypersensitivity reactions

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2015-02; Primary Completion 2016-06 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Safety (adverse events) | 12 weeks after first administration
  Safety assessments will be reported all along the study. The data safety monitoring board will assess Safety at 3 weeks and 12 weeks of treatment.

SECONDARY OUTCOMES:
Efficacy 9 Efficacious dose at 3 weeks will be considered if normalisation of body temperature and decrease of C-reactive protein (CRP) by more or equal to 50 percent of baseline values are achieved.) | 12 weeks after first administration
  Efficacy is assessed by the principal investigator. Efficacious dose at 3 weeks will be considered if normalisation of body temperature and decrease of C-reactive protein (CRP) by more or equal to 50 percent of baseline values are achieved.
  At twelve weeks, the dose will be considered efficacious if normalisation of body temperature persists, and improvement in joint tenderness or swelling (more or equal to 20 percent) and a decrease of CRP and ferritin to reference values.

CONTACTS AND LOCATIONS:
Overall Officials: Cem Gabay, Prof., Principal Investigator — Hospital University of Geneva
Locations (20):
- France (7):
  - Hôpital Pellegrin, Bordeaux
  - CHRU de Lille - Hôpital Claude Huriez, Lille
  - Hôpital de la Croix Rousse, Lyon
  - CHRU de Montpellier, Montpellier
  - CHU de Nantes - Hôtel Dieu, Nantes
  - CHU Paris-GH La Pitié Salpêtrière-Charles Foix - Hôpital Pitié-Salpêtrière, Paris
  - Strasbourg University Hospital, Strasbourg
- Germany (10):
  - Innere Medizin II - Rheumatologie Schlosspark-Klinik, Berlin
  - Medizinische Klinik - Rheumatologie und Klinische, Berlin
  - Universitätsklinikum Erlangen, Erlangen
  - Asklepios Klinik Altona, Hamburg
  - St. Elisabeth Gruppe GmbH Katholische Kliniken Rhein-Ruhr Rheumazentrum Ruhrgebiet, Herne
  - Universitätsklinikum Jena Klinik für Innere Medizin III Rheumatologie/Osteologie, Jena
  - Klinik Kirchheim, Kirchheim unter Teck
  - Universitätsklinikum Schleswig-Holstein - Campus Lübeck, Lübeck
  - UNIVERSITÄTSMEDIZIN der Johannes-Gutenberg-Universität Mainz I. Medizinische Klinik und Poliklinik Rheumatologie, Mainz
  - LMU München, München
- Switzerland (3):
  - Hôpitaux Universitaires de Genève - HUG, Geneva
  - CHUV hospital, Lausanne
  - Immunologie-Zentrum de Zürich, Zurich

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bagnari V, Colina M, Ciancio G, Govoni M, Trotta F. Adult-onset Still's disease. Rheumatol Int. 2010 May;30(7):855-62. doi: 10.1007/s00296-009-1291-y. Epub 2009 Dec 18. PMID 20020138
- [Background] Bywaters EG. Still's disease in the adult. Ann Rheum Dis. 1971 Mar;30(2):121-33. doi: 10.1136/ard.30.2.121. No abstract available. PMID 5315135
- [Background] Efthimiou P, Kontzias A, Ward CM, Ogden NS. Adult-onset Still's disease: can recent advances in our understanding of its pathogenesis lead to targeted therapy? Nat Clin Pract Rheumatol. 2007 Jun;3(6):328-35. doi: 10.1038/ncprheum0510. PMID 17538564
- [Background] Fautrel B. Adult-onset Still disease. Best Pract Res Clin Rheumatol. 2008 Oct;22(5):773-92. doi: 10.1016/j.berh.2008.08.006. PMID 19028363
- [Background] Kawashima M, Yamamura M, Taniai M, Yamauchi H, Tanimoto T, Kurimoto M, Miyawaki S, Amano T, Takeuchi T, Makino H. Levels of interleukin-18 and its binding inhibitors in the blood circulation of patients with adult-onset Still's disease. Arthritis Rheum. 2001 Mar;44(3):550-60. doi: 10.1002/1529-0131(200103)44:33.0.CO;2-5. PMID 11263769
- [Background] Yamaguchi M, Ohta A, Tsunematsu T, Kasukawa R, Mizushima Y, Kashiwagi H, Kashiwazaki S, Tanimoto K, Matsumoto Y, Ota T, et al. Preliminary criteria for classification of adult Still's disease. J Rheumatol. 1992 Mar;19(3):424-30. PMID 1578458
- [Derived] Gabay C, Fautrel B, Rech J, Spertini F, Feist E, Kotter I, Hachulla E, Morel J, Schaeverbeke T, Hamidou MA, Martin T, Hellmich B, Lamprecht P, Schulze-Koops H, Courvoisier DS, Sleight A, Schiffrin EJ. Open-label, multicentre, dose-escalating phase II clinical trial on the safety and efficacy of tadekinig alfa (IL-18BP) in adult-onset Still's disease. Ann Rheum Dis. 2018 Jun;77(6):840-847. doi: 10.1136/annrheumdis-2017-212608. Epub 2018 Feb 22. PMID 29472362